CLINICAL TRIAL: NCT00058669
Title: CVD Risk Factors and Sexual Identity in Women
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nina Markovic, Assoc Professor of Dental Public Health, University of Pittsburgh
Other Study IDs: 1210; R01HL067052 (NIH)
Record Dates: First submitted 2003-04-10; First posted 2003-04-11 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — urine, plasma,
Oversight: Data Monitoring Committee: No

SUMMARY:
To examine potential differences in the prevalence and pattern of risk factors for coronary heart disease in a sample of 500 self-identified lesbians and 500 heterosexual women, matched for age, socioeconomic status, and ethnicity.

DETAILED DESCRIPTION:
BACKGROUND:

Coronary heart disease (CHD) is the leading cause of mortality among women living in the United States, regardless of race and ethnicity and is likely the leading cause of mortality among lesbians. However, in various reports since 1994, the National Institute of Mental Health, the Centers for Disease Control and Prevention, the American Medical Association, the American Public Health Association, and the Institute of Medicine (IOM) have pointed out that health care and health research affecting lesbian women are inadequate. As women, lesbians share many of the same health concerns of all women. However, as emphasized in the IOM Report on Lesbian Health "factors assumed to place women at risk for or to protect them against health disorders may not be present at the same levels or operate in the same way for lesbians". The IOM report also recognizes that "women who self-identify as lesbian may also experience stressors not commonly faced by heterosexual women" and that "it is important to understand the factors that are unique to lesbians and their impact on lesbians' health". Data which do exist from household surveys and studies utilizing convenience samples indicate that women who identify as lesbian may differ from heterosexual women in several important factors which contribute to the development of CHD. However, to date there has not been a comprehensive examination of CHD risk in a large sample of women who identify as lesbian or an examination of how their pattern of risk factors or overall risk for CHD may differ from a sample of demographically similar heterosexual women.

DESIGN NARRATIVE:

The study is a case-control, cross-sectional survey that includes both behavior (alcohol, smoking, substance use, physical activity) and physiological (lipids, blood pressure, adiposity) measures. Self-identified lesbian women will be age, education, and racially matched to heterosexual women. The study will test the hypotheses that the prevalence and pattern of coronary heart disease (CHD) risk factors are different between lesbians and heterosexual women. The study will also determine the absolute and relative risk estimates for CHD based on the Framingham multiple-risk-factor assessment equations, and test the hypothesis that lesbians are at increased risk of CHD compared to heterosexual women.

ELIGIBILITY:
Over 35 Years old no cvd

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women over 35 Years age without cvd
Sampling Method: Non-Probability Sample
Enrollment: 1174 (Actual)
Dates: Start 2003-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
risk of cardiovascular disease | single visit
  Framingham risk profile

CONTACTS AND LOCATIONS:
Overall Officials: nina markovivc, phd, Principal Investigator — University of Pittsburgh